CLINICAL TRIAL: NCT05221320
Title: A Phase 2 Basket Trial of Ulixertinib (BVD-523) in Combination With Hydroxychloroquine in Patients With Advanced GI Malignancies Harboring Mitogen-activated Protein Kinase (MAPK) Pathway Mutations (BVD-523-HCQ)
Brief Title: Trial of Ulixertinib in Combination With Hydroxychloroquine in Patients With Advanced Gastrointestinal (GI) Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment for Remaining Open Baskets
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BVD-523-HCQ
Record Dates: First submitted 2021-12-20; First posted 2022-02-02 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Tumor, Solid; Gastrointestinal Cancer
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms | interventions — ulixertinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage 1 - 5 baskets included, based on primary disease (Experimental): Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
  Interventions: Drug: Ulixertinib; Drug: Hydroxychloroquine
- Stage 2 - basket expansion based on Stage 1 (Experimental): Ulixertinib: 450mg BID, orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
  Interventions: Drug: Ulixertinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Ulixertinib — small molecule ERK 1/2 inhibitor
  Other Names: BVD-523; BVD523
Drug: Hydroxychloroquine — Autophagy inhibitor

SUMMARY:
This is an open-label, prospective phase two basket trial assessing the efficacy of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies. All patients enrolled must have a mitogen-activated protein kinase (MAPK) activating mutation to be deemed eligible for trial participation. Each disease-based basket will open to enrollment in two-stages. The opening of stage two will be dependent on the observed responses in the patients enrolled in the first stage.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II basket study of ulixertinib in combination with hydroxychloroquine in patients with advanced gastrointestinal malignancies harboring rat sarcoma virus (RAS), a member of the rapidly accelerated fibrosarcoma (non-V600 BRAF), extracellular signal-regulated kinase (ERK), or mitogen-activated protein kinase (MEK) mutations. The trial will have five baskets based on disease primary as listed below.

Basket 1: Cholangiocarcinoma including intrahepatic cholangiocarcinoma, perihilar cholangiocarcinoma, or extrahepatic cholangiocarcinoma;

Basket 2: Pancreatic adenocarcinoma;

Basket 3: Colorectal adenocarcinoma;

Basket 4: Esophageal adenocarcinoma, esophageal squamous cell carcinoma, or gastroesophageal junction (GEJ) adenocarcinoma;

Basket 5: Gastric adenocarcinoma.

While the overall trial is a basket design, each basket will operate as a Simon two-stage design and therefore, will open to enrollment in two-stages.

Total enrollment for Stage 1 is targeted at approximately 65 patients with 13 patients per group. Additional patients may be enrolled as appropriate.

Total enrollment for Stage 2 is targeted to approximately 150 patients with up to 30 patients per group. Additional patients may be enrolled as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged ≥ 18 years.
2. Histologically confirmed esophageal adenocarcinoma, esophageal squamous cell carcinoma, GEJ adenocarcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma, intrahepatic cholangiocarcinoma, perihilar cholangiocarcinoma, extrahepatic cholangiocarcinoma, or colorectal adenocarcinoma harboring a MAPK-mutated GI malignancy: KRAS, NRAS, HRAS, BRAF non-V600, MEK 1/2 (MAP2K1/2), or ERK 1/2 (MAPK3/1).
3. Progression on or during standard lines of therapy:

   * Patients with intrahepatic cholangiocarcinoma, perihilar cholangiocarcinoma, or extrahepatic cholangiocarcinoma must have progressed during or after receiving a first-line regimen of gemcitabine/cisplatin unless deemed ineligible by the treating investigator to receive chemotherapy-based regimens due to prior comorbidities.
   * Patients with pancreatic adenocarcinoma must have progressed during or after first-line therapy of FOLFIRINOX/ mFOLFIRINOX, gemcitabine/nab-paclitaxel unless deemed ineligible by the treating investigator to receive chemotherapy-based regimens due to prior comorbidities.
   * Patients with colorectal adenocarcinoma must have progressed during or after their first two lines of therapy, including FOLFOX ± Avastin and FOLFIRI ± Avastin, unless deemed ineligible by the treating investigator to receive chemotherapy-based regimens due to prior comorbidities.
   * Patients with esophageal adenocarcinoma, esophageal squamous cell carcinoma, GEJ adenocarcinoma, or gastric adenocarcinoma must have progressed during or after their first two lines of therapy.
   * Acceptable first-line regimens: FOLFOX, 5-FU/Cisplatin, FOLFIRI, Paclitaxel/Cisplatin or Carboplatin, Docetaxel/Cisplatin, DCF (or modifications thereof), or ECF (or modifications thereof) unless deemed ineligible by the treating investigator to receive chemotherapy-based regimens due to prior comorbidities.
   * Acceptable second-line regimens: Ramucirumab/Paclitaxel, Docetaxel, Paclitaxel, Irinotecan, Trifluridine/Tipiracil, or FOLFIRI, unless deemed ineligible by the treating investigator to receive chemotherapy-based regimens due to prior comorbidities.
   * Patients with deficient MisMatch Repair/High levels of MicroSatellite Instability (dMMR/MSI-H) tumors must have progressed during or after pembrolizumab.
4. Measurable disease by RECIST 1.1 criteria by computed tomography (CT) or magnetic resonance imaging (MRI).
5. Willing to provide a biopsy at the time points indicated on the Schedule of Activities.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
7. Adequate organ function as defined as:

   Hematologic:
   * Absolute neutrophil count (ANC) ≥ 1500/mm3
   * Platelet count ≥ 100,000/mm3
   * Hemoglobin ≥ 9 g/dL

   Hepatic:
   * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
   * Asparate animotransferace /Alanine aminotransferase (AST(SGOT)/ALT(SGPT)) ≤ 3 × institutional ULN
   * Patients with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.

   Renal:
   * Estimated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula:
   * Males:

     (140-age) × weight [kg] / serum creatinine [mgdL] × 72
   * Females:

   ((140-age) × weight [kg] / serum creatinine [mgdL] × 72)×0.85
8. For female patients: Negative serum pregnancy test within 72 hours prior to first dose of study drugs for women of childbearing potential. The following definitions apply:

   * Women of childbearing potential, defined as a sexually mature woman:
   * Has not been naturally post-menopausal for at least 12 consecutive months (i.e., who has had menses anytime in the preceding 12 consecutive months).
   * Has not undergone menopause, surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women not of childbearing potential:
   * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, if any.
   * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. Male and female patients of childbearing potential agree to use highly effective contraception throughout the study and at least 90 days after the last study treatment administration.
10. Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior cancer therapy, unless considered clinically not significant by the treating investigator.
11. Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

1. Received systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any investigational therapy ≤ 14 days or within five half-lives prior to starting study treatment, whichever is shorter.
2. Received radiotherapy ≤ 14 days prior to the first dose of study treatment.

   Note: Localized radiation therapy for the treatment of symptomatic bone metastasis is allowed during that timeframe.
3. Undergone major surgery ≤ 3 weeks prior to starting study drug or who have not fully recovered from major surgery.
4. The diagnosis of another malignancy within ≤ 3 years before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration (i.e., basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, or low-grade prostate cancer with Gleason Score ≤ 6).
5. Known uncontrolled brain metastases or cranial epidural disease.

   Note: Patients with stable brain metastases either treated or being treated with a stable dose of steroids (<20 mg of prednisone daily or equivalent) or anticonvulsants, with no dose change within 4 weeks before the first study drug dose, and no anticipated dose change, are eligible. In the event of steroid taper post-radiation therapy, taper must be complete within 2 weeks before Baseline.
6. History or current evidence of central serous retinopathy (CSR) or retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity).
7. Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

   Cardiovascular disorders:
   * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
   * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 3 months before the first dose.
   * Duration of QT interval (QTc prolongation) defined as a QTcF > 500 ms.
   * Known congenital long QT.
   * Left ventricular ejection fraction < 50%.

   History of seizures

   Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).

   Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [patients may not receive the drug through a feeding tube], social/ psychological issues, etc.)
8. Prior stomach or duodenal resection that in the opinion of the Principal Investigator and Medical Monitor would affect the breakdown and absorption of the study medications. A patient with a feeding tube should also be excluded, as ulixertinib capsules cannot be broken apart.
9. Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

   Note: Patients on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
10. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

    Note: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
11. Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.
12. Known prior severe hypersensitivity to investigational product (IP) or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
13. Patients taking prohibited medications as described in protocol. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Kansas Cancer Center, Fairway, Kansas
  - Rogel Cancer Center, University of Michigan Health, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Massey Cancer Center, Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 sites in the USA. Enrollment took place between May 2022 and July 2024.
Groups:
- Basket 1: Cholangiocarcinoma Including Intrahepatic, Perihilar, Extrahepatic Cholangiocarcinoma; Basket 2 - Pancreatic Adenocarcinoma; Basket 3 - Colorectal Adenocarcinoma; Basket 4 - Esophageal Adenocarcinoma, Esophageal Squamous Cell Gastroesophageal Junction Adeno; Basket 5 - Gastric Adenocarcinoma: Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Basket 1: Cholangiocarcinoma Including Intrahepatic, Perihilar, Extrahepatic Cholangiocarcinoma | Basket 2 - Pancreatic Adenocarcinoma | Basket 3 - Colorectal Adenocarcinoma | Basket 4 - Esophageal Adenocarcinoma, Esophageal Squamous Cell Gastroesophageal Junction Adeno | Basket 5 - Gastric Adenocarcinoma | Stage 2 - Basket Expansion Based on Stage 1
Started | 4 | 18 | 22 | 2 | 1 | 0 (Stage 2 was never started due to trial termination in Stage 1.)
Completed | 0 | 3 | 2 | 0 | 0 | 0
Not Completed | 4 | 15 | 20 | 2 | 1 | 0
Not completed — Lack of Efficacy | 3 | 7 | 10 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 5 | 6 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Stage 2 was never started due to termination in Stage 1.
Groups:
- Basket 2: Pancreatic Adenocarcinoma; Basket 3: Colorectal Adenocarcinoma; Basket 4: Esophageal Adenocarcinoma, Esophageal Squamous Cell, Gastroesophageal Junction; Basket 5: Gastric Adenocarcinoma: Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
- Total: Total of all reporting groups
Arm/Group | Basket 1: Cholangiocarcinoma Including Intrahepatic, Perihilar, Extrahepatic Cholangiocarcinoma | Basket 2: Pancreatic Adenocarcinoma | Basket 3: Colorectal Adenocarcinoma | Basket 4: Esophageal Adenocarcinoma, Esophageal Squamous Cell, Gastroesophageal Junction | Basket 5: Gastric Adenocarcinoma | Stage 2 - Basket Expansion Based on Stage 1 | Total
Number analyzed (Participants) | 4 | 18 | 22 | 2 | 1 | 0 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 10 | 17 | 2 | 0 | 0 | 30
  >=65 years | 3 | 8 | 5 | 0 | 1 | 0 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (14.17) | 62.2 (8.53) | 57.0 (10.76) | 58.5 (6.36) | 68.0 |  | 59.7 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 7 | 0 | 0 | 0 | 18
  Male | 2 | 9 | 15 | 2 | 1 | 0 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 17 | 19 | 2 | 1 | 0 | 43
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 0 | 0 | 4
  White | 3 | 14 | 19 | 2 | 1 | 0 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 18 | 22 | 2 | 1 | 0 | 47
ECOG Performance at Baseline [Count of Participants; unit: Participants] — Measure Description: ECOG performance status was assessed by the clinical site investigator/physician or their designee; ECOG 0 - Fully active, able to carry on all pre-disease performance without restriction; ECOG 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; ECOG 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  Participants
    ECOG 0 | 1 | 5 | 11 | 0 | 0 | 0 | 17
    ECOG 1 | 3 | 13 | 10 | 2 | 1 | 0 | 29
    ECOG 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Smoking History [Count of Participants; unit: Participants]
  Yes - Current Smoker | 0 | 3 | 1 | 1 | 0 | 0 | 5
  Yes - Former | 1 | 5 | 9 | 1 | 0 | 0 | 16
  No - never smoked | 3 | 10 | 12 | 0 | 1 | 0 | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate as Defined by the Proportion of Patients Achieving a Confirmed Partial Response (PR) and Complete Response (CR) (Defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as Evaluated by the Local Treating Investigator.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: from cycle 1 day 1 until safety follow-up visit (up to 24 months)
Population: Outcomes for stage 1 are presented for the total of 47 participants and not broken down by individual basket. None of the patients in Stage 1 met the CR or PR criteria. Stage 2 was never started due to termination of study in Stage 1.
Measure: Count of Participants; unit: Participants
Groups:
- Basket 4 - Esophageal Adenocarcinoma, Esophageal Squamous, Gastroesophageal Junction; Basket 5 - Gastric Adenocarcinoma: Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
Arm/Group | Basket 1: Cholangiocarcinoma Including Intrahepatic, Perihilar, Extrahepatic Cholangiocarcinoma | Basket 2 - Pancreatic Adenocarcinoma | Basket 3 - Colorectal Adenocarcinoma | Basket 4 - Esophageal Adenocarcinoma, Esophageal Squamous, Gastroesophageal Junction | Basket 5 - Gastric Adenocarcinoma | Stage 2 - Basket Expansion Based on Stage 1
Number analyzed (Participants) | 4 | 18 | 22 | 2 | 1 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: The Incidence and Frequency of Serious Adverse Events (SAEs) Characterized by Type, Severity (as Defined by the NCI CTCAE, Version 5.0), Seriousness, Duration, and Relationship to Study Treatment.
Description: Reporting of any SAEs, all SAEs were collected/assessed at each study visit.
Time Frame: Baseline until safety follow-up visit (up to 24 months)
Population: Stage 2 is zero because study was terminated in stage 1.
Measure: Number; unit: Participants
Groups:
- Basket 4 - Esophageal Adenocarcinoma, Esophageal Squamous Cell, Gastroesophageal Junction; Basket 5 - Gastric Adenocarcinoma: Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
Arm/Group | Basket 1: Cholangiocarcinoma Including Intrahepatic, Perihilar, Extrahepatic Cholangiocarcinoma | Basket 2 - Pancreatic Adenocarcinoma | Basket 3 - Colorectal Adenocarcinoma | Basket 4 - Esophageal Adenocarcinoma, Esophageal Squamous Cell, Gastroesophageal Junction | Basket 5 - Gastric Adenocarcinoma | Stage 2 - Basket Expansion Based on Stage 1
Number analyzed (Participants) | 4 | 18 | 22 | 2 | 1 | 0
Participants | 3 | 10 | 12 | 0 | 1 |

3. Primary Outcome: The Incidence and Frequency of Adverse Events (AEs), Characterized by Type, Severity (as Defined by the NCI CTCAE, Version 5.0), Seriousness, Duration, and Relationship to Study Treatment.
Description: Reporting of any AEs, all AEs were collected/assessed at each study visit.
Time Frame: Baseline until safety follow-up visit (up to 24 months)
Population: Stage 2 was never started.
Measure: Number; unit: Participants
Arm/Group | Basket 1: Cholangiocarcinoma Including Intrahepatic, Perihilar, Extrahepatic Cholangiocarcinoma | Basket 2 - Pancreatic Adenocarcinoma | Basket 3 - Colorectal Adenocarcinoma | Basket 4 - Esophageal Adenocarcinoma, Esophageal Squamous Cell, Gastroesophageal Junction | Basket 5 - Gastric Adenocarcinoma | Stage 2 - Basket Expansion Based on Stage 1
Number analyzed (Participants) | 4 | 18 | 22 | 2 | 1 | 0
Participants | 4 | 18 | 22 | 2 | 1 |

4. Secondary Outcome: Progression-free Survival (PFS) as Defined as the Time From Study Drug Initiation to the Time of Documented Disease Progression (as Assessed by RECIST 1.1) or Death From Any Cause.
Description: To assess the duration of efficacy of ulixertinib and hydroxychloroquine in patients with advanced, RAS, non-V600 BRAF, ERK, or MEK mutated gastrointestinal malignancies.
Time Frame: 18 months
Population: Stage 2 is zero because study was terminated in stage 1.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Stage 1 - Cholangiocarcinoma: Basket 1: Cholangiocarcinoma including intrahepatic, perihilar, or extrahepatic cholangiocarcinoma
  Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
- Stage 1 - Pancreas: Basket 2: Pancreatic adenocarcinoma
  Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
- Stage 1 - Colorectal: Basket 3: Colorectal adenocarcinoma
  Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
- Stage 1 - Esophageal: Basket 4: Esophageal adenocarcinoma, esophageal squamous cell carcinoma, or gastroesophageal junction adenocarcinoma
  Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
- Stage 1 - Gastric: Basket 5: Gastric adenocarcinoma
  Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
Arm/Group | Stage 1 - Cholangiocarcinoma | Stage 1 - Pancreas | Stage 1 - Colorectal | Stage 1 - Esophageal | Stage 1 - Gastric | Stage 2 - Basket Expansion Based on Stage 1
Number analyzed (Participants) | 2 | 16 | 22 | 2 | 1 | 0
months | 5.5 [0.7 to 5.5] | 1.9 [1.7 to 2.1] | 1.8 [1.4 to 1.8] | 2.8 [1.7 to 3.9] | 0.7 [0.7 to 0.7] |

ADVERSE EVENTS:
Time Frame: All reportable events were recorded with start dates occurring any time after informed consent obtained through and including 30 calendar days after the last administration of ulixertinib and hydroxychloroquine. The median (min; max) number of cycles received was 2 (1; 6). The median (min; max) duration of exposure was 1.74 (0.0; 5.5) months. All patients fell well within the estimated 24 months.
Description: If there is more than one medical history within a system organ class (SOC), the patient is counted only once under that SOC. If there is more than one medical history within a SOC and preferred term (PT), the patient is counted only once in that SOC and PT.
  AEs were collected/assessed at each study visit.
Groups:
- Stage 1 - Cholangiocarcinoma: Ulixertinib: 450mg twice daily (BID), orally, days 1-28
  Hydroxychloroquine: 600mg BID, orally, days 1-28
  Cycles repeat every 28 days in absence of disease progression or unacceptable toxicity
Arm/Group | Stage 1 - Cholangiocarcinoma | Stage 1 - Pancreas | Stage 1 - Colorectal | Stage 1 - Esophageal | Stage 1 - Gastric | Stage 2 - Basket Expansion Based on Stage 1
All-Cause Mortality (participants affected / at risk) | 1/4 | 12/18 | 15/22 | 2/2 | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/4 | 10/18 | 12/22 | 0/2 | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 18/18 | 22/22 | 2/2 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 - Cholangiocarcinoma (N=4) | Stage 1 - Pancreas (N=18) | Stage 1 - Colorectal (N=22) | Stage 1 - Esophageal (N=2) | Stage 1 - Gastric (N=1) | Stage 2 - Basket Expansion Based on Stage 1 (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Disease progression (General disorders) | 0 (0) | 7 (7) | 5 (5) | 0 (0) | 0 (0) | 0
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Biliary obstruction (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 - Cholangiocarcinoma (N=4) | Stage 1 - Pancreas (N=18) | Stage 1 - Colorectal (N=22) | Stage 1 - Esophageal (N=2) | Stage 1 - Gastric (N=1) | Stage 2 - Basket Expansion Based on Stage 1 (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 14 (14) | 2 (2) | 0 (0) | 0
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (8) | 10 (10) | 0 (0) | 0 (0) | 0
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (7) | 5 (5) | 0 (0) | 0 (0) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 8 (8) | 0 (0) | 0 (0) | 0
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | NA
Dyspepsis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Fatigue (General disorders) | 1 (1) | 7 (7) | 12 (12) | 0 (0) | 1 (1) | 0
Disease Progression (General disorders) | 0 (0) | 7 (7) | 5 (5) | 0 (0) | 0 (0) | 0
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 9 (9) | 0 (0) | 0 (0) | 0
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 0
Weight decreased (Investigations) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0
Protein total decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 9 (9) | 8 (8) | 1 (1) | 0 (0) | 0
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0
Hypocalcaemia (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0
Hypophosphataemia (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 | 0
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0

LIMITATIONS AND CAVEATS:
Baskets 2 and 3 did not proceed past stage 1 due to futility. No definite conclusions can be drawn from baskets 1, 4 and 5 due to slow enrollment and early closure of the study.

Early termination leading to small numbers of patients analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT05221320/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05221320/SAP_001.pdf